CLINICAL TRIAL: NCT00368108
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy, Safety, and Tolerability of E2007 in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Brief Title: Efficacy, Safety, and Tolerability of E2007 in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2007-A001-302
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 2 mg perampanel (Experimental): The Perampanel 2mg dosage was fixed for the entire double-blind study. Subjects taking perampanel 2mg were to take the dose orally once every day in the evening.
  Interventions: Drug: 2 mg perampanel
- 4 mg perampanel (Experimental): The Perampanel 4mg group first were subjected to a 4 week titration period, followed by a maintenance period for the remaining weeks. Subjects taking perampanel 4mg had a titration period of 4 weeks, starting at 2mg per day adding 1mg of perampel every two weeks up to 4mg. The dosages were to be taken orally once every day in the evening.
  Interventions: Drug: 4 mg perampanel
- placebo (Placebo Comparator): The placebo dosage was a fixed dosage for the entire double-blind study. Subjects receiving the placebo were to take one dose orally once every day in the evening.
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: 2 mg perampanel — 2 mg perampanel
  Arms: 2 mg perampanel
Drug: 4 mg perampanel — 4 mg perampanel
  Arms: 4 mg perampanel
Drug: placebo comparator — placebo comparator
  Arms: placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel-group study of E2007 in levodopa treated Parkinson's disease patients with motor fluctuations.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female patients with idiopathic Parkinson's Disease fulfilling the United Kingdom (UK) Parkinson's disease Society Brain Bank diagnostic criteria 7, with a good response to levodopa.
2. Patients must have been diagnosed with idiopathic PD at > 30 years of age.
3. Patients must have predictable motor fluctuations of the wearing "OFF" type.
4. Patients must rate between II-IV on the Hoehn & Yahr scale when in an "OFF" state.
5. Patients must be taking optimized levodopa therapy.

EXCLUSION CRITERIA:

1. Pregnant or lactating women.
2. Women of child bearing potential unless infertile (including surgically sterile) or practicing effective contraception (eg, abstinence, intrauterine device or barrier method plus hormonal method). These patients must have a negative serum beta-human chorionic gonadotrophin (B-HCG) test at the Screening visit, and a negative urine pregnancy test at the Baseline visit (Day 0). These patients must also be willing to remain on their current form of contraception for the duration of the study. Postmenopausal women may be recruited but must be amenorrheic for at least one year to be considered of non-child bearing potential as determined by the Investigator.
3. Patients with a past or present history of drug or alcohol abuse as per Diagnostic and Statistical Manual - 4th edition (DSM IV) criteria.
4. Patients with a past (within one year) or present history of suicidal ideation or suicide attempts.
5. Patients with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, gastro-intestinal, hematological, endocrine or metabolic systems which might complicate assessment of the tolerability of the study medication.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, M.D., Study Director — Eisai Inc.
Locations (114):
- United States (99):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - North Alabama Neuroscience Research Associates, Huntsville, Alabama
  - Pivotal Research Centers, Peoria, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - Clinical Trials Inc., Little Rock, Arkansas
  - UAMS Department of Neurology, Little Rock, Arkansas
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Margolin Brain Institute, Fresno, California
  - University of California Medical Center - Irvine, Irvine, California
  - Coastal Neurological Group, La Jolla, California
  - Scripps Clinic, La Jolla, California
  - University of California at San Diego - Department of Neurology, La Jolla, California
  - Loma Linda University, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - Pacific Neuroscience Medical Group, Inc., Oxnard, California
  - University of California San Francisco Medical Center, San Francisco, California
  - The Parkinson's Institute, Sunnyvale, California
  - Mile High Research Center, Denver, Colorado
  - University Of Colorado, Denver, Colorado
  - Colorado Neurology, Englewood, Colorado
  - Associated Neurologists, PC - Danbury, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Molecular Neuroimaging, LLC, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - University of Florida, Gainesville, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - University of Florida - Department of Neurology, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Miami Research Associates, Miami, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Gil, Ramon A., Port Charlotte, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - University Of South Florida Movement Disorders Clinic, Tampa, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Dekalb Neurology Associates, LLC/DNA Research, Decatur, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University, Indianapolis, Indiana
  - University Of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - University Of Kentucky, Lexington, Kentucky
  - Kentucky Neuroscience Research, Louisville, Kentucky
  - LSUHSC-Shreveport, Shreveport, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Parkinson's and Movement Disorders Center of Maryland, Elkridge, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Quest Research Institute, Bingham Farms, Michigan
  - The Clinical Neurosciences Center, Southfield, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Creighton University - Department of Neurology, Omaha, Nebraska
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - Parkinson's Disease and Movement Disorder Center of Long Island, Commack, New York
  - New York University Medical Center, Forest Hills, New York
  - North Shore Medical Center, Manhasset, New York
  - The Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester - Neurology Clinic, Rochester, New York
  - Asheville Neurology Specialists. PA, Asheville, North Carolina
  - Asheville Neurology Specialists, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Neurology Specialists, Inc., Dayton, Ohio
  - The University of Toledo College of Medicine, Toledo, Ohio
  - University of Oklahoma - Health Sciences Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Crozer Medical Center, Upland, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Semmes Murphey Neurology and Spine Institute, Memphis, Tennessee
  - Radiant Research - Dallas North, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Agape' Medical Center, Inc., Lubbock, Texas
  - Bhupesh Dihenia, MD, PA, Lubbock, Texas
  - Neurology Associates, San Antonio, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Hunter Holmes McGuire, Richmond, Virginia
  - Neurology and Neurosurgery Associates of Tacoma, PLLC, Tacoma, Washington
  - Capitol Neurology, Charleston, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Wisconsin Institute for Neurologic and Sleep Disorders, Milwaukee, Wisconsin
- Canada (15):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Pacific Parkinson Research Centre, Vancouver, British Columbia
  - Saint John Regional Hospital, 5DN, Saint John, New Brunswick
  - David King, MD, Halifax, Nova Scotia
  - Centre For Movement Disorders, Markham, Ontario
  - Parkinson's and Neurodegenerative Disorders Clinic, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Torotnto Western Hospital-University Health Network, Toronto, Ontario
  - Clinique Neuro Rive-Sud, Greenfield Park, Quebec
  - CHUM- Hotel-Dieu, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - SMBD Jewish General Hospital, Montreal, Quebec
  - Quebec Memory and Motor Skills Disorders Clinic, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel 2mg: The Perampanel 2mg dosage was fixed for the entire double-blind study. Subjects taking perampanel 2mg were to take the dose orally once every day in the evening.
- Perampanel 4mg: The Perampanel 4mg group first were subjected to a 4 week titration period, followed by a maintenance period for the remaining weeks. Subjects taking perampanel 4mg had a titration period of 4 weeks, starting at 2mg per day adding 1mg of perampanel every two weeks up to 4mg. The dosages were to be taken orally once every day in the evening.
Period: Overall Study
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg
Started | 251 (One subject had stopped medication prior to notifying staff. Remaining results will have 250.) | 251 | 250
Completed | 187 | 198 | 182
Not Completed | 64 | 53 | 68
Not completed — Adverse Event | 38 | 26 | 44
Not completed — Abnormal Laboratory Value | 0 | 0 | 3
Not completed — Protocol Violation | 5 | 9 | 9
Not completed — Withdrawal by Subject | 9 | 3 | 5
Not completed — Lack of Efficacy | 7 | 8 | 5
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Other | 3 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Total
Number analyzed (Participants) | 250 | 251 | 250 | 751
Age, Customized [Number; unit: Participants]
  <65 years | 149 | 144 | 147 | 440
  ≥ 65 years | 101 | 107 | 103 | 311
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 87 | 86 | 259
  Male | 164 | 164 | 164 | 492
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 233 | 239 | 240 | 712
  Black | 4 | 2 | 1 | 7
  Asian | 5 | 4 | 1 | 10
  Other | 8 | 6 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Daily OFF Time (Hours) to Week 20 (Including Last Observation Carried Forward [LOCF] Data)
Description: Patients described themselves in home diaries as "OFF", "ON" without dyskinesias, "ON" with non troublesome dyskinesias, "ON" with troublesome dyskinesias, or Asleep, every 30 minutes during waking hours for 3 consecutive days prior to Baseline, Weeks 8, 10, 18, and 20. OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline and Week 20
Population: The Intent-to-treat (ITT) Population for diary data consisted of all subjects who were randomized to either perampanel or placebo, had taken at least 1 dose, had a valid, nonmissing Baseline diary measurement and at least 1 valid, non-missing, postbaseline diary measurement at Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg
Number analyzed (Participants) | 208 | 213 | 201
Hours | -0.96 [-1.42 to -0.51] | -0.93 [-1.38 to -0.49] | -0.76 [-1.20 to -0.31]

2. Secondary Outcome: Mean Change From Baseline in Scale UPDRS Part II (ADL) Score in Total Daily OFF Time to Week 20 (Including LOCF Data)
Description: Patients described themselves in home diaries every 30 minutes during waking hours for 3 consecutive days prior to Baseline, Weeks 8, 12, 16, and 20. Unified Parkinson's Disease (PD) Rating Scale (UPDRS) is a standardized assessment of the symptoms and signs of PD. Part II assesses Activities of Daily Living (ADL) based on 13 items, such as speech, hygiene, and falling. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. Range of possible total scores, 0 to 52. ON state is when medication is providing benefits to mobility, slowness, and stiffness. OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline and Week 20
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg
Number analyzed (Participants) | 213 | 216 | 211
Scores on a scale | -0.85 [-1.70 to -0.00] | -0.81 [-1.66 to 0.04] | -1.40 [-2.23 to -0.56]

3. Secondary Outcome: Mean Change From Baseline in UPDRS Part III (Motor) Score in ON State (Hours) to Week 20 (Including LOCF Data)
Description: Patients described themselves in home diaries every 30 minutes during waking hours for 3 days prior to Baseline, Weeks 8, 12, 16, and 20. UPDRS is a standardized assessment of the symptoms and signs of PD. Part III assesses motor activity, based on 14 items, such as gait, facial expression, and rigidity. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. ON state is when medication is providing benefits to stiffness, slowness, and tremor.
Time Frame: Baseline and Week 20
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg
Number analyzed (Participants) | 213 | 215 | 210
Scores on a Scale | -2.15 [-3.59 to -0.71] | -1.69 [-3.13 to -0.25] | -3.29 [-4.71 to -1.87]

4. Secondary Outcome: Mean Change From Baseline in Total Daily ON Time (Without Dyskinesias or With Non-troublesome Dyskinesias) (Hours) to Week 20 (Including LOCF Data)
Description: Patients described themselves in home diaries every 30 minutes during waking hours for 3 days prior to Baseline, Weeks 8, 12, 16, and 20. ON state is when medication is providing benefits to stiffness, slowness, and tremor.
Time Frame: Baseline and Week 20
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg
Number analyzed (Participants) | 208 | 213 | 201
Hours | 0.73 [0.29 to 1.18] | 0.78 [0.33 to 1.22] | 0.28 [-0.15 to 0.72]

ADVERSE EVENTS:
Time Frame: From the time the subject signed the informed consent form to 30 days after the last dose of the study drug.
Description: Adverse events were assessed at clinical visits based on the subject's diary, vitals, weight, physical examination, neurological exam, and laboratory evaluations.
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg
Serious Adverse Events (participants affected / at risk) | 22/250 | 12/251 | 18/250
Other Adverse Events (participants affected / at risk) | 111/250 | 110/251 | 144/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=250) | Perampanel 2mg (N=251) | Perampanel 4mg (N=250)
Syncope (Nervous system disorders) | 1 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1
ON and OFF phenomenon (Nervous system disorders) | 0 | 1 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 | 0 | 0
Tonic convulsion (Nervous system disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Cardio-Respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hospitalization (Surgical and medical procedures) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=250) | Perampanel 2mg (N=251) | Perampanel 4mg (N=250)
Nausea (Gastrointestinal disorders) | 16 | 11 | 12
Urinary Tract Infection (Infections and infestations) | 10 | 11 | 13
Fall (Injury, poisoning and procedural complications) | 23 | 23 | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 16 | 12
Balance Disorder (Nervous system disorders) | 3 | 6 | 17
Dizziness (Nervous system disorders) | 14 | 15 | 29
Dyskinesia (Nervous system disorders) | 39 | 21 | 43
Headache (Nervous system disorders) | 18 | 10 | 12
ON and OFF phenomenon (Nervous system disorders) | 24 | 18 | 21
Somnolence (Nervous system disorders) | 13 | 32 | 40
Insomnia (Psychiatric disorders) | 15 | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No